CLINICAL TRIAL: NCT01147406
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single-Dose Escalation Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effect of N6022 in Healthy Subjects
Brief Title: Safety and Tolerability Study of N6022 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nivalis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N6022-1H1-01
Record Dates: First submitted 2010-06-14; First posted 2010-06-22 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
MeSH Terms: interventions — N6022

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): N6022
  Interventions: Drug: N6022
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N6022 — This is an injectible formulation which will be given at 5, 15 & 45 mg over 1, 3 and 9 minutes respectively, in single ascending doses.
  Arms: Active
Drug: Placebo — This will be 0.9% normal saline given over 1, 3, or 9 minutes IV bolus.
  Other Names: N6022
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of N6022 in healthy subjects.

DETAILED DESCRIPTION:
This is a single dose escalation, first-time-in-human study with three ascending cohorts. Eligible subjects will receive a single dose of investigational medicinal product or placebo on Day 1 and will be followed for safety, PK, and PD for 72 hours post dose. Follow-up visits on Day 4 and Day 7 for the end-of-study safety. Participation of an individual subject may last up to 36 days from the time of screening until the end-of-study follow-up visit. Each cohort will enroll a sentinel pair (1:1 randomized to active: placebo). These subjects will be followed for 48 hours postdose and safety data reviewed before the remaining subjects in the cohort receive IMP. A Safety Monitoring Committee will review the seven-day safety data in each cohort before proceeding to the next ascending dose cohort, according to the stopping rules outlined in the protocol.

ELIGIBILITY:
Inclusion:

* Subject is healthy

Exclusion:

* Subject is a current alcohol abuser and/or has a history of illicit drug abuse within six months of entry.
* Subject has donated blood (> 500 mL) or blood products within 56 days prior to Day -1

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, MDCM, MSc(A), Principal Investigator — Parexel
Locations (1):
- Parexel Early Phase Unit, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 5 mg of N6022 was given intravenously daily for 7 days
- Cohorts 2 and 4: 15 mg of N6022 was given intravenously daily for 7 days
- Cohort 3: 45 mg of N6022 was to be given intravenously daily for 7 days however, the actual amount was 27.5 mg.
- Cohort 5: 25 mg of N6022 was given intravenously daily for 7 days
- Cohort 6: 35 mg of N6022 was given intravenously daily for 7 days
- Placebo: Not Active - Placebo
Period: Overall Study
Arm/Group | Cohort 1 | Cohorts 2 and 4 | Cohort 3 | Cohort 5 | Cohort 6 | Placebo
Started | 6 | 12 | 1 | 6 | 6 | 10
Completed | 6 | 12 | 1 | 6 | 6 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Any subject that received any active or placebo
Groups:
- Cohort 1: N6022 - Active 5 mg
- Cohort 2 & 4: N6022 - Active 15 mg
- Cohort 3: N6022 - Active 45 mg (actual *27.5 mg)
- Cohort 5: N6022 - Active 25 mg
- Cohort 6: N6022 - Active 35 mg
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 & 4 | Cohort 3 | Cohort 5 | Cohort 6 | Placebo | Total
Number analyzed (Participants) | 6 | 12 | 1 | 6 | 6 | 10 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 12 | 1 | 6 | 6 | 10 | 41
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 12 | 1 | 6 | 6 | 10 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 9 | 1 | 4 | 5 | 6 | 30
  White | 1 | 3 | 0 | 2 | 1 | 4 | 11
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 6 | 12 | 1 | 5 | 6 | 9 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 12 | 1 | 6 | 6 | 10 | 41

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of a Single Ascending Doses of Intravenous N6022 in Healthy Volunteers
Description: Safety variables - number of adverse events reported during study, changes in vital signs, physical examination findings, telemetry alerts, 12-lead ECG changes, infusion site reactions, O2 saturation changes, and clinical laboratory assessment changes between subjects receiving N6022 versus placebo.
Time Frame: 7 Days
Population: Any subject that received active IMP or placebo
Measure: Number; unit: Adverse Events
Groups:
- Cohort 2 and 4: N6022 - Active 15 mg
- Cohort 3: N6022 - Active 45 mg
Arm/Group | Cohort 1 | Cohort 2 and 4 | Cohort 3 | Cohort 5 | Cohort 6 | Placebo
Number analyzed (Participants) | 6 | 12 | 1 | 6 | 6 | 10
Adverse Events | 1 | 4 | 1 | 0 | 1 | 2

2. Secondary Outcome: Maximum N6022 and Metabolite Concentrations in Plasma Within 24 Hours of End of Administration
Description: Concentrations of N6022 and metabolite [N61149)], collected on Days 1 and 7; predose, end of infusion, and at 10 minutes, 30 minutes, 1, 2, 4, 6, 8, 12, 16, and 24 hours post-dose (the 24 hour postdose collected prior to the start of infusion on Day 2).
Time Frame: 24 hours
Population: Any subject that received the active IMP or placebo
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2 and 4 | Cohort 3 | Cohort 5 | Cohort 6 | Placebo
Number analyzed (Participants) | 6 | 12 | 1 | 6 | 6 | 10
ng/mL | 311 (86.6) | 1570 (51.5) | 1590 (0) | 3330 (42.1) | 4030 (55.3) | 0 (0)

ADVERSE EVENTS:
Time Frame: 6 months and 2 weeks
Arm/Group | Cohort 1 | Cohort 2 and 4 | Cohort 3 | Cohort 5 | Cohort 6 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/12 | 0/1 | 0/6 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 1/6 | 4/12 | 1/1 | 0/6 | 1/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6) | Cohort 2 and 4 (N=12) | Cohort 3 (N=1) | Cohort 5 (N=6) | Cohort 6 (N=6) | Placebo (N=6)
Injection Site Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — and administration site conditions
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection Site Hematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — and administration site conditions
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — administration and site conditions
Sinus Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees with the use of results of the clinical study for the purposes of national and international registration, publication, and information for medical and pharmaceutical professionals. If necessary, the competent authorities will be notified of the investigator's name, address, qualifications, and extent of involvement. An investigator shall not publish any data (poster, abstract, paper, etc.) without having consulted with the Sponsor in advance.